CLINICAL TRIAL: NCT04495127
Title: A Phase 1 Open Label Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of Selumetinib, a Selective Mitogen Activated Protein Kinase Kinase (MEK) 1 Inhibitor, in Japanese Paediatric Subjects With Neurofibromatosis Type 1 (NF1) and Inoperable and Symptomatic Plexiform Neurofibromas (PN)
Brief Title: Selumetinib Paediatric NF1 Japan Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1346C00013
Record Dates: First submitted 2020-07-29; First posted 2020-07-31 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — AZD 6244

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selumetinib (Experimental)
  Interventions: Drug: Selumetinib

INTERVENTIONS:
Drug: Selumetinib — Selumetinib 25 mg/m2 BID

SUMMARY:
This is a phase I open label study designed to evaluate the safety, tolerability, PK and efficacy of selumetinib in Japanese paediatric patients with neurofibromatosis type 1 and inoperable and symptomatic plexiform neurofibroma.

ELIGIBILITY:
Key Inclusion Criteria:

* Three years of age or older, and less than or equal to 18 years of age at the time of obtaining informed consent. BSA greater than or equal to 0.55 m2, and able to swallow the whole study drug (capsules) without entire contents unpacked from the capsules.
* NF1 and inoperable and symptomatic PN who have PN-related morbidities (symptom and/or complications), as judged by the investigator.
* Inoperable PN is defined as PN that cannot be surgically completely removed without risk for substantial morbidity due to encasement of, or close proximity to, vital structures, invasiveness, or high vascularity of the PN.
* A PN is defined as a neurofibroma that has grown along the length of a nerve and may involve multiple fascicles and branches. A spinal PN involves two or more levels with connection between the levels or extending laterally along the nerve.
* In addition to PN, subjects must have at least 1 other diagnostic criterion for NF1 as follows:

  1. Six or more café-au-lait macules >5 mm in greatest diameter in pre-pubertal individuals and >15 mm in greatest diameter in post-pubertal individuals.
  2. Freckling in the axillary or inguinal regions.
  3. Optic glioma.
  4. Two or more Lisch nodules (iris hamartomas).
  5. A distinctive osseous lesion such as sphenoid dysplasia or tibial pseudarthrosis.
  6. A first-degree relative with NF1.
* At least one measurable typical or nodular PN in principle, defined as a lesion of at least 3 cm measured in one dimension.
* Adequate organ/haematological function

Key Exclusion Criteria:

* Evidence of malignant peripheral nerve sheath tumour.
* Prior malignancy (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, low grade optic pathway gliomas associated with NF1 which does not require systemic treatment or other cancer from which the subject had been disease free for ≥2 years or which would not have limited survival to <2 years) or other cancer requiring treatment with chemotherapy or radiation therapy.
* Clinically significant cardiovascular disease
* Known history of human immunodeficiency virus, serologic status reflecting active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, or any uncontrolled active systemic infection
* Subjects with clinically significant ophthalmological findings/conditions
* Inability to undergo MRI and/or contraindication for MRI (i.e. prosthesis or orthopaedic or dental braces that would interfere with volumetric analysis of target PN on MRI).
* Have refractory nausea and vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease), or significant bowel resection that would adversely affect the absorption/bioavailability of the orally administered study medication.
* Receiving supplementation with vitamin E greater than 100% of the daily recommended dose.
* Receiving herbal supplements or medications known to be strong inhibitors or inducers of the cytochrome P450 (CYP) 3A4 enzymes unless such products can be safely discontinued at least 14 days before the first dose of study medication.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability in terms of adverse events | From obtaining the first informed consent until 30 days after the last dose (Selumetinib). Expected duration is approximately 2 years.
  Number of subjects with adverse events as a measure of safety and tolerability including changes in vital signs, electrocardiograms, safety laboratory parameters, echocardiogram and ophthalmologic assessment.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | From obtaining the first informed consent until 30 days after the last dose (Selumetinib). Expected duration is approximately two years.
  Pharmacokinetics (PK) parameters will be derived using standard non-compartmental methods.
Area under the plasma concentration-time curve (AUC) | From obtaining the first informed consent until 30 days after the last dose (Selumetinib). Expected duration is approximately two years.
  Pharmacokinetics (PK) parameters will be derived using standard non-compartmental methods.
Overall response rate | Assessed at every 4 cycles until drug permanently discontinued. Expected duration is approximately 2 years. Each cycle is 28 days.
  Defined as the proportion of subjects who achieve a response by independent central review per Response Evaluation in Neurofibromatosis and Schwannomatosis (REiNS) criteria.
Duration of response | Assessed at every 4 cycles until drug permanently discontinued. Expected duration is approximately 2 years. Each cycle is 28 days.
  Defined as the time from the date of the first documented response (which is subsequently confirmed) until the date of documented progression or death in the absence of disease progression, as determined by independent central review per REiNS criteria.
Clinical Global Impression of Change (CGIC) | Assessed at every 2 cycles for the first year and every 4 cycles until drug permanently discontinued. Expected duration is approximately 2 years. Each cycle is 28 days.
  Comprehensive evaluation will be performed by investigator on the changes of PN related morbidities (symptoms and/or complications), and relevant findings including imaging studies and physical exams from baseline.
Total scale score of Paediatric Quality of Life Inventory (PedsQL; self- and parent-reported) | Assessed at every 4 cycles until drug permanently discontinued. Expected duration is approximately 2 years. Each cycle is 28 days.
  Scale scores are computed as the sum of the items divided by the number of items answered (this accounts for missing data). A Total Scale Score will also be derived as the sum of all the items divided by the number of items answered on all the scales.

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Research Site, Minatoku
  - Research Site, Nagoya
  - Research Site, Setagaya-ku

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home